CLINICAL TRIAL: NCT04401696
Title: Comparison of Bubble Nasal Continuous Positive Airway Pressure (bCPAP) Versus Control in Neonates With Respiratory Distress
Brief Title: Effectiveness of Bubble Nasal Continuous Positive Airway Pressure (bCPAP) in Neonatal Respiratory Distress
Acronym: bCPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Tehreem Fatima, Tehreem Fatima, Senior Registrar, Children Hospital & ICH Faisalabad., King Edward Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BubbleCPAP
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Neonatal Respiratory Distress
Keywords: bubble CPAP; respiratory distress; neonates; Silverman Anderson Retraction Score
MeSH Terms: conditions — Pulmonary Atelectasis; Dyspnea

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Use of Bubble CPAP for management of respiratory distress
  Interventions: Device: Bubble CPAP
- Group B (Active Comparator): Use of Oxygen via nasal cannula for respiratory distress
  Interventions: Other: Nasal Oxygen

INTERVENTIONS:
Device: Bubble CPAP — The bCPAP will be delivered using an oxygen flow meter as the oxygen source. This inspiratory limb containing oxygen from the flow meter will be connected to humidifier and tubing from humidifier will be connected to short binasal prongs, which would be applied to neonate with the help of adhesive bandage on both cheeks. It will be ensured that binasal prongs make appropriate seal. An orogastric tube will be placed for gastric decompression. A 1000 ml/500ml bottle filled with sterile water be used and marks will be made on it at 1cm distance, with '10' marked at base and '0' mark at the water interface.
  The expiratory limb from the nasal prongs was connected to tubing that will be dipped in water up to the desired level to provide positive end expiratory pressure. Pressure is varied by varying the depth of the dipped end of tubing.
  Arms: Group A
Other: Nasal Oxygen — The oxygen will be delivered from a wall oxygen source, delivered between 1 to 6 L/min and the rate varied via a flow regulator.
  Arms: Group B

SUMMARY:
The objective of study is to determine the effectiveness of bubble Continuous Positive Airway Pressure (bCPAP) in neonates presenting with respiratory distress as compared to the control group ( using oxygen via nasal cannula). The effectiveness will be calculated in terms of reduction in Silverman Anderson Retraction Score.

DETAILED DESCRIPTION:
After approval from the IRB of King Edward Medical University, and taking informed consent from parents of the participants, total of 120 neonates fulfilling inclusion and exclusion criteria will be enrolled and randomly allocated in two groups; group A and group B. All demographic details of participants in both groups be collected. In group A, neonates will be given bCPAP for respiratory support while neonates in group B, will be given nasal oxygen as control group. Neonates in both groups will be followed for 48 hours. The effectiveness will be determined by the reduction in Silverman Anderson Retraction Score (SARS) up to or less than 3, at the end of 48 hours. Data will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients having age 28 days of life or younger (Neonates)
* Gender- both male and female
* Gestational ages ≥32 weeks
* Having respiratory distress (as per the operational definition- respiratory rate >60/min plus any of the following features: grunting, subcostal/intercostal retractions, nasal flaring, inability to maintain spO2 >90% at room air)
* Silverman Anderson Retraction Score ≥4

Exclusion Criteria:

* Neonates having gestational age less than 32 weeks
* Birth weight less than 1.5 kg
* Neonates having congenital malformations, air leak syndromes, hypoxic ischemic encephalopathy
* Neonates requiring mechanical ventilation at the time of admission

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Bubble CPAP determined by improvement in Silvermann Anderson Retraction Score | 48 hours since application of intervention
  Neonates in both groups will be followed-up for 48 hours. SAR Score will be recorded at 0 and 48 hours. It consists of five components: (1) chest retractions (2) retraction of the lower intercostal muscles (3) xiphoid retractions (4) flaring of nares with inhalation (5) grunting on exhalation. Each of the five factors is graded 0, 1 and 2. The sum of these factors yields the total score; minimum score is '0' and maximum score is '10'. The higher the score, the greater is the severity of respiratory distress. So the severity of respiratory distress can be graded according to the SAR Score as Mild (score 0-3), Moderate (score4-6) and Severe (score 6-10). Effectiveness is recorded as 'positive' in case of reduction in SARS score ≤3. A cut-off of score '3' is taken. So if the score of 3 or less than 3 is achieved with bCPAP or with nasal oxygen after 48 hours of intervention, the intervention is considered to be effective

SECONDARY OUTCOMES:
Mean reduction in SAR Score | 48 hours
  Mean reduction in Silverman Anderson Retraction Score, over a period of 48 hours, in both groups
Difference in mean reduction | 48 hours
  difference between both the groups, will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Tehreem Fatima, FCPS, Principal Investigator — King Edward Medical University
Locations (1):
- King Edward Medical University/ Mayo Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen A, Deshmukh AA, Richards-Kortum R, Molyneux E, Kawaza K, Cantor SB. Cost-effectiveness analysis of a low-cost bubble CPAP device in providing ventilatory support for neonates in Malawi - a preliminary report. BMC Pediatr. 2014 Nov 25;14:288. doi: 10.1186/s12887-014-0288-1. PMID 25421903
- [Background] Mustufa MA, Korejo R, Shahid A, Nasim S. Infection remains a leading cause of neonatal mortality among infants delivered at a tertiary hospital in Karachi, Pakistan. J Infect Dev Ctries. 2014 Sep 13;8(11):1470-5. doi: 10.3855/jidc.3569. PMID 25390060
- [Background] Daga S, Mhatre S, Borhade A, Khan D. Home-made continuous positive airways pressure device may reduce mortality in neonates with respiratory distress in low-resource setting. J Trop Pediatr. 2014 Oct;60(5):343-7. doi: 10.1093/tropej/fmu023. Epub 2014 Apr 23. PMID 24760748
- [Background] Kawaza K, Machen HE, Brown J, Mwanza Z, Iniguez S, Gest A, Smith EO, Oden M, Richards-Kortum RR, Molyneux E. Efficacy of a low-cost bubble CPAP system in treatment of respiratory distress in a neonatal ward in Malawi. PLoS One. 2014 Jan 29;9(1):e86327. doi: 10.1371/journal.pone.0086327. eCollection 2014. PMID 24489715
- [Background] Brown J, Machen H, Kawaza K, Mwanza Z, Iniguez S, Lang H, Gest A, Kennedy N, Miros R, Richards-Kortum R, Molyneux E, Oden M. A high-value, low-cost bubble continuous positive airway pressure system for low-resource settings: technical assessment and initial case reports. PLoS One. 2013;8(1):e53622. doi: 10.1371/journal.pone.0053622. Epub 2013 Jan 23. PMID 23372661
- [Background] Stoll BJ, Hansen NI, Bell EF, Walsh MC, Carlo WA, Shankaran S, Laptook AR, Sanchez PJ, Van Meurs KP, Wyckoff M, Das A, Hale EC, Ball MB, Newman NS, Schibler K, Poindexter BB, Kennedy KA, Cotten CM, Watterberg KL, D'Angio CT, DeMauro SB, Truog WE, Devaskar U, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Trends in Care Practices, Morbidity, and Mortality of Extremely Preterm Neonates, 1993-2012. JAMA. 2015 Sep 8;314(10):1039-51. doi: 10.1001/jama.2015.10244. PMID 26348753
- [Background] Hundalani SG, Richards-Kortum R, Oden M, Kawaza K, Gest A, Molyneux E. Development and validation of a simple algorithm for initiation of CPAP in neonates with respiratory distress in Malawi. Arch Dis Child Fetal Neonatal Ed. 2015 Jul;100(4):F332-6. doi: 10.1136/archdischild-2014-308082. Epub 2015 Apr 15. PMID 25877290
- [Background] Kaur C, Sema A, Beri RS, Puliyel JM. A simple circuit to deliver bubbling CPAP. Indian Pediatr. 2008 Apr;45(4):312-4. PMID 18451452
- [Background] Anwaar O, Hussain M, Shakeel M, Ahsan Baig MM. Outcome Of Use Of Nasal Continuous Positive Airway Pressure Through Infant Flow Drivers In Neonates With Respiratory Distress In A Tertiary Care Hospital In Pakistan. J Ayub Med Coll Abbottabad. 2018 Oct-Dec;30(4):511-555. PMID 30632326
- [Background] Hedstrom AB, Gove NE, Mayock DE, Batra M. Performance of the Silverman Andersen Respiratory Severity Score in predicting PCO2 and respiratory support in newborns: a prospective cohort study. J Perinatol. 2018 May;38(5):505-511. doi: 10.1038/s41372-018-0049-3. Epub 2018 Feb 9. PMID 29426853
- [Background] Wilson PT, Baiden F, Brooks JC, Morris MC, Giessler K, Punguyire D, Apio G, Agyeman-Ampromfi A, Lopez-Pintado S, Sylverken J, Nyarko-Jectey K, Tagbor H, Moresky RT. Continuous positive airway pressure for children with undifferentiated respiratory distress in Ghana: an open-label, cluster, crossover trial. Lancet Glob Health. 2017 Jun;5(6):e615-e623. doi: 10.1016/S2214-109X(17)30145-6. PMID 28495265
- [Background] Al-Lawama M, Alkhatib H, Wakileh Z, Elqaisi R, AlMassad G, Badran E, Hartman T. Bubble CPAP therapy for neonatal respiratory distress in level III neonatal unit in Amman, Jordan: a prospective observational study. Int J Gen Med. 2018 Dec 24;12:25-30. doi: 10.2147/IJGM.S185264. eCollection 2019. PMID 30636889